CLINICAL TRIAL: NCT02278263
Title: Tranexamic Acid in Knee Joint Surgery - a Randomised Controlled Trial
Brief Title: Tranexamic Acid in Knee Joint Surgery
Acronym: TRACKS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andrew G Hill, MBChB, MD (Thesis), EdD, FACS, FRACS (Other)
Responsible Party: Sponsor-Investigator, Andrew G Hill, MBChB, MD (Thesis), EdD, FACS, FRACS, Professor of Surgery, University of Auckland, New Zealand
Organization: University of Auckland, New Zealand (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRACKS Study
Record Dates: First submitted 2014-09-18; First posted 2014-10-29 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Osteoarthritis
Keywords: tranexamic acid; enhanced recovery; arthroplasty; perioperative care
MeSH Terms: conditions — Osteoarthritis | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Application of 20ml of normal saline (NaCl 0.9%) topically after implantation of prosthesis and left to sit for two minutes, excess carefully suctioned followed by standard closure with no drains; application of 15ml of normal saline intravenously at the same time prior to release of tourniquet.
  Interventions: Drug: Normal saline (0.9% NaCl)
- Topical (Experimental): Application of 1.5g in 20ml tranexamic acid topically after implantation of prosthesis with excess carefully suctioned followed by standard closure with no drains; application of 15ml of normal saline intravenously at the same time prior to release of tourniquet.
  Interventions: Drug: Tranexamic Acid; Drug: Normal saline (0.9% NaCl)
- Systemic (Experimental): Application of 20ml of normal saline topically after implantation of prosthesis with excess carefully suctioned followed by standard closure with no drains; Application of tranexamic acid intravenously (1.5g/15ml) at the same time prior to release of tourniquet
  Interventions: Drug: Tranexamic Acid; Drug: Normal saline (0.9% NaCl)

INTERVENTIONS:
Drug: Tranexamic Acid — Given intravenously or topically
  Other Names: Cyclokapron
  Arms: Systemic; Topical
Drug: Normal saline (0.9% NaCl) — Administered in all 3 groups
  Other Names: Normal saline

SUMMARY:
Total knee joint replacement surgery can lead to significant blood loss, which can affect recovery after surgery. Tranexamic acid (TXA) is a medication which stops the breakdown of blood clots and therefore prevents blood loss. The optimal use of TXA remains a point of debate. Growing interest in the topical application of TXA (directly into the surgical wound) has been suggested as an alternative way of administering TXA, and may demonstrate similar effectiveness as when it is given intravenously. Therefore, this multicentred, randomized controlled trial, aims to investigate the safety and effectiveness of both topical and intravenous administrations of TXA in total knee joint surgery. The investigators predict that both routes of administration will demonstrate similar results when compared to placebo.

DETAILED DESCRIPTION:
Postoperative anaemia following elective arthroplasty can lead to prolonged hospital stay, delays in rehabilitation and is often poorly tolerated in patients with cardiovascular disease.(1) Tranexamic acid (TXA) in arthroplasty is used by many orthopaedic surgeons to reduce perioperative blood loss and subsequent transfusion of blood products in elective total hip and knee arthroplasty (THA and TKA). In several reviews, systemic TXA (sTXA) significantly reduces blood loss and transfusion rates when compared to placebo, without an increased risk for venous thromboembolism (VTE).(2-4)

The CRASH-2 study, with over 20,000 randomised trauma patients, has also confirmed the efficacy and safety of TXA in this setting, particularly when given early.(5) The evidence for its use to date is overwhelming and when not contraindicated, should be employed by all arthroplasty units as part of their standard practice. However, despite the vast evidence for its use in arthroplasty some surgeons remain cautious over its safety profile when given systemically. TXA is a synthetic derivative of lysine which is responsible for binding reversibly to plasminogen effectively inhibiting clot degradation.(6) Although, this is not clot promoting, inhibiting clot breakdown theoretically may increase the likelihood of clot formation. This is of real concern for surgeons in patients who have had previous VTE. For this reason, some surgeons have utilised TXA as a topical application directly into the surgical field to reduce systemic absorption and avoid VTE.(7, 8)

TXA administered topically in TKA has also been reported to reduce swelling which may have the advantage of earlier mobility and less pain.(9) In cardiac surgery, TXA has been touted as not only having blood conserving properties via the coagulation pathway but also reduces inflammation via attenuation of the pro-inflammatory cascade.(10, 11)

Based on this rationale, this appears to be a sensible and reasonable route of administration for TXA in this population. However, surgeons should ensure they avoid placing undue risk on patients by altering their use of TXA given the strong evidence for sTXA. Therefore, the purpose of this study is to assess whether topical TXA is effective in reducing blood loss in knee joint replacement surgery, and is as safe and as effective as systemic TXA.

ELIGIBILITY:
Inclusion Criteria:

* All patients at the participating sites on the waiting list for a unilateral total knee joint replacement

Exclusion Criteria:

* Patients with a history or risk of thrombosis
* Active thromboembolic disease such as deep vein thrombosis, pulmonary embolism and cerebral thrombosis
* Subarachnoid haemorrhage
* Hypersensitivity to tranexamic acid or any of its ingredients.
* Refusal of blood products
* Colour blindness
* Complex hematologic disorders requiring manipulation
* Coagulopathy
* Pregnant and Lactating Women
* Anti-coagulant therapy pre-operatively within 5 days of surgery (warfarin, dabigatran, heparin)
* Severe renal failure (eGFR <29)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob T Munro, MBChB, FRACS, Principal Investigator — Department of Surgery, The University of Auckland
Locations (5):
- New Zealand (5):
  - Auckland Hospital, Auckland
  - Manukau Surgery Centre, Auckland
  - North Shore Hospital, Auckland
  - Nelson Hospital, Nelson
  - Tauranga Hospital, Tauranga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carson JL, Duff A, Berlin JA, Lawrence VA, Poses RM, Huber EC, O'Hara DA, Noveck H, Strom BL. Perioperative blood transfusion and postoperative mortality. JAMA. 1998 Jan 21;279(3):199-205. doi: 10.1001/jama.279.3.199. PMID 9438739
- [Background] Alshryda S, Sarda P, Sukeik M, Nargol A, Blenkinsopp J, Mason JM. Tranexamic acid in total knee replacement: a systematic review and meta-analysis. J Bone Joint Surg Br. 2011 Dec;93(12):1577-85. doi: 10.1302/0301-620X.93B12.26989. PMID 22161917
- [Background] Sukeik M, Alshryda S, Haddad FS, Mason JM. Systematic review and meta-analysis of the use of tranexamic acid in total hip replacement. J Bone Joint Surg Br. 2011 Jan;93(1):39-46. doi: 10.1302/0301-620X.93B1.24984. PMID 21196541
- [Background] Gandhi R, Evans HM, Mahomed SR, Mahomed NN. Tranexamic acid and the reduction of blood loss in total knee and hip arthroplasty: a meta-analysis. BMC Res Notes. 2013 May 7;6:184. doi: 10.1186/1756-0500-6-184. PMID 23651507
- [Background] CRASH-2 collaborators; Roberts I, Shakur H, Afolabi A, Brohi K, Coats T, Dewan Y, Gando S, Guyatt G, Hunt BJ, Morales C, Perel P, Prieto-Merino D, Woolley T. The importance of early treatment with tranexamic acid in bleeding trauma patients: an exploratory analysis of the CRASH-2 randomised controlled trial. Lancet. 2011 Mar 26;377(9771):1096-101, 1101.e1-2. doi: 10.1016/S0140-6736(11)60278-X. PMID 21439633
- [Background] Williams-Johnson JA, McDonald AH, Strachan GG, Williams EW. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2) A randomised, placebo-controlled trial. West Indian Med J. 2010 Dec;59(6):612-24. PMID 21702233
- [Background] Wind TC, Barfield WR, Moskal JT. The effect of tranexamic acid on blood loss and transfusion rate in primary total knee arthroplasty. J Arthroplasty. 2013 Aug;28(7):1080-3. doi: 10.1016/j.arth.2012.11.016. Epub 2013 Mar 28. PMID 23541868
- [Background] Wind TC, Barfield WR, Moskal JT. The effect of tranexamic acid on transfusion rate in primary total hip arthroplasty. J Arthroplasty. 2014 Feb;29(2):387-9. doi: 10.1016/j.arth.2013.05.026. Epub 2013 Jun 21. PMID 23790499
- [Background] Ishida K, Tsumura N, Kitagawa A, Hamamura S, Fukuda K, Dogaki Y, Kubo S, Matsumoto T, Matsushita T, Chin T, Iguchi T, Kurosaka M, Kuroda R. Intra-articular injection of tranexamic acid reduces not only blood loss but also knee joint swelling after total knee arthroplasty. Int Orthop. 2011 Nov;35(11):1639-45. doi: 10.1007/s00264-010-1205-3. Epub 2011 Jan 21. PMID 21253725
- [Background] Later AF, Sitniakowsky LS, van Hilten JA, van de Watering L, Brand A, Smit NP, Klautz RJ. Antifibrinolytics attenuate inflammatory gene expression after cardiac surgery. J Thorac Cardiovasc Surg. 2013 Jun;145(6):1611-6, 1616.e1-4. doi: 10.1016/j.jtcvs.2012.11.042. Epub 2013 Jan 16. PMID 23332183
- [Background] Robertshaw HJ. An anti-inflammatory role for tranexamic acid in cardiac surgery? Crit Care. 2008;12(1):105. doi: 10.1186/cc6210. Epub 2008 Jan 16. PMID 18254939
- [Derived] Stowers MDJ, Aoina J, Vane A, Poutawera V, Hill AG, Munro JT. Tranexamic Acid in Knee Surgery Study-A Multicentered, Randomized, Controlled Trial. J Arthroplasty. 2017 Nov;32(11):3379-3384. doi: 10.1016/j.arth.2017.05.058. Epub 2017 Jun 9. PMID 28662956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The hospital databases will be searched for eligible patients on the waiting list for unilateral total knee joint replacement. Patients will be approached in the preadmission clinics and then consented on the day of surgery. Recruitment period is to be over 2 years or sooner once we have recruited the final patient (n=150)
Pre-assignment Details: Patients were excluded after consenting to participate, if they failed to receive spinal anaesthesia.
Groups:
- Control: Application of 20ml of normal saline (NaCl 0.9%) topically after implantation of prosthesis; application of 15ml of normal saline intravenously at the same time prior to release of tourniquet.
  Normal saline (0.9% NaCl): Administered in all 3 groups
- Intraarticular: Application of 1.5g in 20ml tranexamic acid topically after implantation of prosthesis; application of 15ml of normal saline intravenously at the same time prior to release of tourniquet.
  Tranexamic Acid: Given intraarticularly
  Normal saline (0.9% NaCl): Administered in all 3 groups
- Systemic: Application of 20ml of normal saline topically after implantation of prosthesis; Application of tranexamic acid intravenously (1.5g/15ml) at the same time prior to release of tourniquet
  Tranexamic Acid: Given intravenously
  Normal saline (0.9% NaCl): Administered in all 3 groups
Period: Overall Study
Arm/Group | Control | Intraarticular | Systemic
Started | 30 | 60 | 60
Completed | 23 | 60 (Correction) | 51
Not Completed | 7 | 0 | 9
Not completed — Protocol Violation | 7 | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intraarticular | Systemic | Total
Number analyzed (Participants) | 23 | 60 | 51 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 15 | 11 | 32
  >=65 years | 17 | 45 | 40 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.67 (7.75) | 69.72 (8.85) | 70.79 (8.61) | 70.12 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 32 | 24 | 75
  Male | 4 | 28 | 27 | 59
Region of Enrollment [Number; unit: participants]
  New Zealand | 23 | 60 | 51 | 134
Preoperative Hb [Mean (Standard Deviation); unit: grams/L] | 134 (11.8) | 138 (12.2) | 138 (10.6) | 137 (11.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.3 (6.6) | 31.2 (5.5) | 31.2 (5.5) | 31.3 (5.7)
Preop Hb (number of days prior to surgery date) [Mean (Standard Deviation); unit: days] | 28 (34) | 39 (40) | 28 (34) | 31 (33)

OUTCOME MEASURES:

1. Primary Outcome: Blood Loss
Description: The loss of haemoglobin (Hb) was then estimated according to the formula:
  Hb(loss) = Blood volume (BV) x (Hbi-Hbe) x 0.001+Hbt
  where Hb (loss) (g) is the amount of Hb lost, Hbi (g/L) the Hb concentration before surgery, Hbe (g/L) is the Hbe concentration on the third day after surgery, and Hbt (g) is the total amount of allogeneic Hb transfused. A unit of banked blood is considered to contain a minimum of 40g Hb (Blood component data sheet, New Zealand Blood Services [NZBS]). All units of blood are processed and stored in a nationally standardised manner. The blood loss (ml) was related to the patient's preoperative Hb value (g/L):
  Blood loss =1000 x Hb(loss) /Hbi
Time Frame: Post operative day 3
Population: The number provided here for each group are those patients analyzed after patients had been excluded due to breaches in the study protocol. As stated in the power calculation for this primary outcome, an attrition rate of 15% (ie breaches in study protocol, drop out etc) had been accounted for. Hence the discrepancy.
Measure: Mean (Standard Deviation); unit: mls
Arm/Group | Control | Intraarticular | Systemic
Number analyzed (Participants) | 23 | 60 | 51
mls | 1090 (589) | 716 (377) | 746 (321)
Statistical Analysis 1: Comparison: Control vs Intraarticular vs Systemic; Assuming a common standard deviation of 412 mL, to detect a difference of 300 mL of blood loss between the two treatment arms (sTXA and tTXA) and the placebo group, a sample size of 125 participants is required for a statistical power of 0.85, and a type I error of 0.05. The sample size required was 125 participants in total. The was increased by 15% to allow for expected dropouts. Therefore, a minimum of 147 patients was required for the study; Test type: Superiority; p < 0.05, ANOVA

2. Secondary Outcome: Number of Participants Experiencing Symptomatic Venothromboembolic (VTE) Disease
Description: Rates of deep vein thrombosis (DVT) and pulmonary embolus (PE) in each group recorded as a percentage
Time Frame: Postoperatively within 30 days after surgery
Population: Logistic regression for categorical/binary outcomes
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Topical | Systemic
Number analyzed (Participants) | 23 | 60 | 51
Participants
  DVT | 0 | 0 | 0
  PE | 0 | 2 | 1

3. Secondary Outcome: Number of Participants Receiving Allogenic Blood Transfusion
Description: Those patients receiving blood products. Standardised protocol is as follows:
  The criterion for transfusion of blood products will be a haemoglobin < 80g/L or a haemoglobin <100g/L in a patient with ischaemic heart disease or with significant symptomatology
Time Frame: Participants will be followed for the duration of their hospital stay expected to be an average of 3-5 days
Population: Logistic regression for binary outcomes
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Topical | Systemic
Number analyzed (Participants) | 23 | 60 | 51
Participants | 2 | 1 | 0

4. Secondary Outcome: Length of Stay (LOS)
Description: Day of surgery is counted as Day 0.
Time Frame: Average length of stay is expected to be 3 to 5 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Topical | Systemic
Number analyzed (Participants) | 23 | 60 | 51
days | 4 [3 to 5] | 4 [3 to 4] | 4 [3 to 5]

5. Secondary Outcome: Range of Passive Flexion
Description: Range of motion measured in degrees for postoperative days 1 to 3
Time Frame: Days 1-3
Population: Range of passive flexion measured and the data presented here are the averages with standard deviations
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control | Topical | Systemic
Number analyzed (Participants) | 23 | 60 | 51
degrees
  Day 1 | 65 (28) | 74 (15) | 68 (15)
  Day 2 | 76 (15) | 81 (13) | 80 (13)
  Day 3 | 82 (13) | 87 (11) | 87 (13)

6. Secondary Outcome: Range of Active Flexion
Description: Range of motion measured in degrees on postoperative days 1-3
Time Frame: Days 1-3
Population: Range of active flexion measured and the data presented here represent the average active flexion with SD.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control | Topical | Systemic
Number analyzed (Participants) | 23 | 60 | 51
degrees
  Day 1 | 57 (23) | 65 (18) | 58 (16)
  Day 2 | 71 (15) | 75 (14) | 72 (16)
  Day 3 | 75 (11) | 82 (12) | 78 (16)

7. Secondary Outcome: Perioperative Fluid Administration
Description: Intravenous fluid (excluding blood transfusion) given during and first 24 hours after surgery
Time Frame: Day 1
Measure: Mean (95% Confidence Interval); unit: mls
Arm/Group | Control | Topical | Systemic
Number analyzed (Participants) | 23 | 60 | 51
mls | 1765 [1320 to 2209] | 1613 [1455 to 1770] | 1807 [1581 to 2033]

ADVERSE EVENTS:
Time Frame: 30 days
Description: The total number at risk is now consistent with the numbers provided in the participant flow module. This also applies to the 'Other adverse events' data table.
Arm/Group | Control | Intraarticular | Systemic
Serious Adverse Events (participants affected / at risk) | 0/23 | 2/60 | 1/51
Other Adverse Events (participants affected / at risk) | 3/23 | 4/60 | 5/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=23) | Intraarticular (N=60) | Systemic (N=51)
Infection (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=23) | Intraarticular (N=60) | Systemic (N=51)
Blood transfusion (Blood and lymphatic system disorders) | 3 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No